CLINICAL TRIAL: NCT05717296
Title: Evaluation of the Effectiveness of a Multimedia Information Site in Reducing Preoperative Anxiety in Vascular Surgery Patients. A Controlled Trial
Brief Title: Evaluation of the Effectiveness of a Multimedia Information Site in Reducing Preoperative Anxiety in Vascular Surgery Patients.
Acronym: VASCUORG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-A00664-39
Record Dates: First submitted 2022-09-20; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-09

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with multimedia support (Experimental)
  Interventions: Other: anxiety survey; Other: scale of satisfaction; Other: Multimedia Information
- without multimedia support (Sham Comparator)
  Interventions: Other: anxiety survey

INTERVENTIONS:
Other: anxiety survey — surgery and anesthesia anxiety questionnaire
Other: scale of satisfaction — scale of satisfaction of multimedia
  Arms: with multimedia support
Other: Multimedia Information — Patients randomized to the "with multimedia support arm "will have access to educational videos focused on the vascular surgery they are to receive.
  Arms: with multimedia support

SUMMARY:
Anxiety is a phenomenon that frequently occurs before surgery. Preoperative anxiety has been studied in several disciplines, including rheumatology, anesthesia, stomatology and cardiology. The implications of preoperative anxiety in terms of morbidity and mortality have also been studied and are well known: intraoperative hemodynamic disorders, increased postoperative mortality, increased consumption of anesthetic agents.

Several scales have been developed to quantify preoperative anxiety, the most frequently used being the visual analog scale and the Amsterdam scale. Several approaches have been considered to reduce preoperative anxiety, such as hypnosis, music, or multimedia.

However, no consensus tool has been developed for vascular surgery patients. Similarly, no study has examined preoperative anxiety in this specific population.

The aim of this study is to evaluate a new multimedia information medium for vascular surgery patients and to assess its effectiveness in reducing preoperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient affiliated to a health insurance plan
* French-speaking patient
* Patient who has given free, informed and express consent
* Patient who has consulted a vascular surgeon for a scheduled procedure
* Patient with internet and telephone access to view videos
* Patient referred for surgical or endovascular treatment for obliterative arteriopathy of the lower limbs, abdominal aortic aneurysm and surgical treatment for carotid stenosis

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patients with blindness
* Patients with severe cognitive impairment
* Patients without access to a digital support to view the videos
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-06-29 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the evolution of preoperative anxiety in patients with access to multimedia with the help of a numerical scale compared to the group of patients without multimedia support | Day 0 ; Day 1 ; Day before the surgery
  The patient rates his anxiety between 0 and 10: 0 no anxiety; 10 maximum anxiety

SECONDARY OUTCOMES:
Assessment of satisfaction with the multimedia support using a 4-point scale: 1) Very satisfied ; 2) Satisfied ; 3) Not very satisfied ; 4) Not satisfied | Day before the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Paris Saint Joseph-hopital Marie Lannelongue, Le Plessis-Robinson, Île-de-France Region, France